CLINICAL TRIAL: NCT04625556
Title: Development of Urologic Registry for Personalized Medicine in Patients With Urologic Malignant Diseases by Analyzing Microbiome
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1018
Record Dates: First submitted 2020-10-29; First posted 2020-11-12 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Urological Malignancies; Prostate Cancer; Renal Cell Cancer; Bladder Cancer; Ureter Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — frozen tissue, blood, stool, and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Prostate cancer: Patients diagnosed as prostate cancer and have undergone prostatectomy
- Renal cell cancer: Patients diagnosed as renal cell cancer and have undergone partial or radical nephrectomy
- Bladder cancer: Patients diagnosed as bladder cancer and have undergone radical or partial cystectomy
- Ureter cancer: Patients diagnosed as ureter cancer and have undergone nephroureterectomy or ureterectomy

SUMMARY:
Genitourinary malignancies such as prostate cancer, renal cell cancer, and bladder cancer in Korean population have been increased due to the aged population and the westernized lifestyles. With the advancement of technologies, studies have found that microbiome not only affects human physiological functions, such as metabolism, immunity, and haematopoiesis, but also plays a significant role in the development and progression of malignancies. However, the investigation of microbiome in urological malignances have been limited and few studies have been reported. Therefore, the investigator tried to evaluate the usefulness of microbiome in detection and monitoring of urological malignancies in Korean population. This study aims to use microbiome in tissue, plasma, stool and urine for the diagnosis, disease progression monitoring and therapeutic response evaluation. This study plan includes building big databases for microbiome of urological malignancies in Korean population.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as urological malignancies (prostate cancer, renal cell cancer, bladder cancer, and ureter cancer)
* Patients who have undergone surgeries due to urological malignancies in Severance Hospital, Sinchon from 2020.10 and 2030.10
* Those who agree to give permission to use their human source information
* Those who agree with this study

Exclusion Criteria:

* Those who do not agree with this study
* Vulnerable participants who are likely to be vulnerable to coercion or undue influence or lack decision-making

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone surgeries with urological malignancies (prostate cancer, renal cell cancer, bladder cancer, and ureter cancer) in Severance Hospital, Sinchon from 2020.10 and 2030.10 were selected.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between tissue bacteria composition and prevalence of urological malignancies | within 2 weeks after the surgery
  evaluate and compare the bacteria composition in tissue samples in urological malignancies (prostate cancer, renal cell cancer, bladder cancer, and ureter cancer) with healthy control group
Correlation between plasma bacteria composition and prevalence of urological malignancies | within 2 weeks after the surgery
  evaluate and compare the bacteria composition in plasma samples in urological malignancies (prostate cancer, renal cell cancer, bladder cancer, and ureter cancer) with healthy control group
Correlation between stool bacteria composition and prevalence of urological malignancies | within 2 weeks after the surgery
  evaluate and compare the bacteria composition in stool samples in urological malignancies (prostate cancer, renal cell cancer, bladder cancer, and ureter cancer) with healthy control group
Correlation between urine bacteria composition and prevalence of urological malignancies | within 2 weeks after the surgery
  evaluate and compare the bacteria composition in urine samples in urological malignancies (prostate cancer, renal cell cancer, bladder cancer, and ureter cancer) with healthy control group

SECONDARY OUTCOMES:
Correlation of bacteria composition and tumor response assessed using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) | within 10 years after the surgery
  Association between bacteria composition and oncological prognosis, progression, and therapeutic response in urological malignancies

CONTACTS AND LOCATIONS:
Overall Officials: Won Sik Ham, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No